CLINICAL TRIAL: NCT02365376
Title: Collection and Storage of Human Biospecimens for Research Into Rare Diseases and Medical Conditions
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: BioMarin Pharmaceutical (Industry)
Responsible Party: Sponsor
Other Study IDs: BMN 000-901
Record Dates: First submitted 2015-02-11; First posted 2015-02-18 (Estimated); Last update posted 2015-02-18 (Estimated); Status verified 2015-02

CONDITIONS: Rare Genetic Disorders

STUDY DESIGN:
Observational Model: Case-Only
Oversight: Data Monitoring Committee: No

SUMMARY:
The objective of this protocol is to enable collection of biospecimens to facilitate current and future multidisciplinary research in rare genetic disorders and medical conditions.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide written, signed informed consent
* Willing and able to comply with all study procedures

Exclusion Criteria:

* Use of any investigational product or investigational medical device within 30 days prior to screening, except as part of a BioMarin-sponsored study
* Concurrent disease or condition that would interfere with study participation or safety.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Individuals diagnosed with rare genetic diseases or medical conditions actively being investigated by BioMarin.
Sampling Method: Non-Probability Sample
Dates: Start 2013-06

PRIMARY OUTCOMES:
continuous collection of donated study subject samples | unknown, continuous sample collection

CONTACTS AND LOCATIONS:
Locations (1):
- Lurie Children's Hospital of Chicago, Chicago, Illinois, United States